CLINICAL TRIAL: NCT03539536
Title: Phase 2, Open-Label Safety and Efficacy Study of Telisotuzumab Vedotin (ABBV-399) in Subjects With Previously Treated c-Met+ Non-Small Cell Lung Cancer
Brief Title: Study of Telisotuzumab Vedotin (ABBV-399) in Participants With Previously Treated c-Met+ Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M14-239; 2023-507902-15-00 (Other: EU CT)
Expanded Access: NCT04830202 (Available)
Record Dates: First submitted 2018-05-17; First posted 2018-05-29 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer (NSCLC); Cancer; Telisotuzumab vedotin; ABBV-399; c-Met, c-Met overexpression; metastatic; MET gene amplification; LUMINOSITY
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis | interventions — telisotuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Telisotuzumab vedotin (Experimental): Telisotuzumab vedotin administered via intravenous (IV) infusion every 14 days.
  Interventions: Drug: Telisotuzumab vedotin

INTERVENTIONS:
Drug: Telisotuzumab vedotin — Intravenous (IV) infusion
  Other Names: ABBV-399

SUMMARY:
This study is designed to identify the target Non-Small Cell Lung Cancer (NSCLC) population(s) that overexpress c-Met (c-Met+) best suited for telisotuzumab vedotin therapy in the second line or third line setting (Stage 1) and then to expand the group(s) to further evaluate efficacy in the selected population(s) (Stage 2). After the Stage 2 global enrollment is completed, an additional cohort at an alternate dose level will evaluate the safety and efficacy of telisotuzumab vedotin (Stage 3).

ELIGIBILITY:
Inclusion Criteria:

* Have locally advanced or metastatic non-small cell lung cancer (NSCLC).
* Have c-Met+ NSCLC as assessed by an AbbVie designated immunohistochemistry (IHC) laboratory. Participant must submit archival or fresh tumor material for assessment of c-Met levels during the prescreening period. Tumor material from the primary tumor site and/or metastatic sites are allowed. If archival tissue is negative for c-Met overexpression, subject can submit fresh biopsy material for reassessment of c-Met expression.
* Histologically documented non-squamous epidermal growth factor receptor (EGFR) wild type NSCLC (site documented EGFR status). Of note, subjects with other actionable mutations are eligible as long as EGFR status is known and all other eligibility criteria are met. As of Protocol Version 11, Stage 1 is complete and Stage 2 is enrolling participants with non-squamous EGFR wild type NSCLC only.
* Must have received no more than 2 lines of prior systemic therapy (including no more than 1 line of systemic cytotoxic chemotherapy) in the locally advanced or metastatic setting.
* Multiple lines of tyrosine kinase inhibitors (TKIs) targeting the same tyrosine kinase (TK) count as 1 line of therapy for the purposes of this eligibility criterion.
* Progressed on systemic cytotoxic therapy (or are ineligible for systemic cytotoxic chemotherapy) and an immune checkpoint inhibitor (as monotherapy or in combination with systemic cytotoxic chemotherapy, or ineligible), and prior anticancer therapies targeting driver gene alterations (if applicable).
* Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1.
* Treatment with any therapies within the noted time intervals is excluded prior to the first dose of telisotuzumab vedotin as noted in the protocol.
* Metastases to the central nervous system (CNS) are eligible only after definitive therapy (such as surgery or radiotherapy) is provided within the protocol.

Exclusion Criteria:

* Have received radiation therapy to the lungs < 6 months prior to the first dose of telisotuzumab vedotin.
* Have received any live vaccine within 30 days of the first dose of investigational product.
* Has adenosquamous histology.
* Have a history of other malignancies except those noted within the protocol.
* Have a history of interstitial lung disease (ILD) or pneumonitis that required treatment with systemic steroids.
* Have any evidence of pulmonary fibrosis on screening imaging assessment or any history of pneumonitis or ILD within 3 months of the planned first dose of the study drug (Except for Sites in Ireland). For imaging findings deemed clinically insignificant by the treating physician, subject may be eligible after discussion with and approval from the AbbVie medical monitor.
* For Sites in Ireland Only: Must not have any evidence of pulmonary fibrosis on screening imaging assessment or any history of pneumonitis or ILD. For imaging findings deemed clinically insignificant by the treating physician, subject may be eligible after discussion with and approval from the AbbVie medical monitor.
* Have a clinically significant condition(s) as noted in the protocol.
* Have unresolved clinically significant adverse events of Grade >= 2 from prior anticancer therapy, except for alopecia or anemia.
* Have had major surgery within 21 days prior to the first dose of telisotuzumab vedotin.
* For Sites in France and Czech Republic Only: Have the following:

  * Known human immunodeficiency virus (HIV) infection. Note: HIV testing is not required for eligibility for this protocol unless mandated by local regulatory authority or ethics committee/institutional review board.
  * Active hepatitis B virus (HBV) infection, defined by hepatitis B surface antigen (HBsAg) positivity or HBV DNA >= 500 IU/mL. In participants with known HBV infection, the presence of active infection must be tested locally. If HBV status is unknown, it must be tested locally at screening.
  * Active hepatitis C virus (HCV) infection, defined by HCV ribonucleic acid (RNA) positivity. Participants cured of HCV infection may be included in the study. In participants with known HCV infection, the presence of active infection must be tested locally. If HCV status is unknown, it must be tested locally at screening.
  * Uncontrolled autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) (Stage 1 and Stage 2) | Up to approximately 3 years
  ORR is defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1.
Number of Participants with Adverse Events (Alternate dose cohort) | Up to approximately 3 years
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Duration of Response (DoR) (Stage 1 and Stage 2) | Up to approximately 3 years
  DoR is defined as the time from the participant's initial response (CR or PR) to the first occurrence of radiographic progression determined by an independent central review or death from any cause for the responders.
Disease Control Rate (DCR) (Stage 1 and Stage 2) | Up to approximately 3 years
  DCR is defined as the percentage of participants with best overall response of confirmed CR, confirmed PR, or stable disease (SD) for at least 12 weeks following enrollment, based on RECIST, version 1.1.
Progression-Free Survival (PFS) (Stage 1 and Stage 2) | Up to approximately 3 years
  PFS is defined as the time from the participant's first dose of study drug until the first occurrence of radiographic progression determined by an independent central review or death from any cause.
Overall Survival (OS) (Stage 1 and Stage 2) | Up to approximately 3 years
  OS is defined as the time from the participant's first dose of study drug until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (252):
- United States (56):
  - University of South Alabama /ID# 212939, Mobile, Alabama
  - Mayo Clinic Arizona /ID# 218550, Phoenix, Arizona
  - Highlands Oncology Group, PA /ID# 215600, Springdale, Arkansas
  - University of California, Los Angeles /ID# 203219, Los Angeles, California
  - LA Hematology-Oncology Med Group /ID# 203338, Orange, California
  - Sutter Medical Center Sacramen /ID# 203299, Sacramento, California
  - Icri /Id# 227835, Whittier, California
  - Univ of Colorado Cancer Center /ID# 203212, Aurora, Colorado
  - Duplicate_Rocky Mountain Cancer Centers - Lone Tree /ID# 215789, Lone Tree, Colorado
  - Advanced Cancer Treatment Center /ID# 239565, Brooksville, Florida
  - AdventHealth Celebration /ID# 215649, Celebration, Florida
  - Duplicate_Mayo Clinic /ID# 218488, Jacksonville, Florida
  - Duplicate_AdventHealth Cancer Institute - Orlando /ID# 239960, Orlando, Florida
  - Straub Clinic and Hospital /ID# 217905, Honolulu, Hawaii
  - Northwestern University Feinberg School of Medicine /ID# 203239, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 203216, Chicago, Illinois
  - Duplicate_NorthShore University HealthSystem /ID# 215583, Evanston, Illinois
  - Ingalls Memorial Hosp /ID# 203228, Harvey, Illinois
  - Joliet Oncology-Hematology Associates, LTD /ID# 203238, Joliet, Illinois
  - Goshen Center for Cancer Care /ID# 215584, Goshen, Indiana
  - Univ Kansas Med Ctr /ID# 216804, Kansas City, Kansas
  - Cancer Center of Kansas /ID# 203235, Wichita, Kansas
  - Duplicate_Baptist Health /ID# 203283, Lexington, Kentucky
  - Duplicate_Norton Cancer Institute - St Matthews /ID# 203284, Louisville, Kentucky
  - Central Maine Medical Center /ID# 216583, Lewiston, Maine
  - Massachusetts General Hospital /ID# 203215, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center /ID# 208124, Boston, Massachusetts
  - Dana-Farber Cancer Institute /ID# 203248, Boston, Massachusetts
  - Henry Ford Hospital /ID# 203220, Detroit, Michigan
  - Mayo Clinic - Rochester /ID# 215603, Rochester, Minnesota
  - Hattiesburg Clinic /ID# 227691, Hattiesburg, Mississippi
  - St. Lukes Cancer Institute /ID# 227697, Kansas City, Missouri
  - Washington University-School of Medicine /ID# 203217, St Louis, Missouri
  - Duplicate_Intermountain Health - St Vincent Regional Hospital - Cancer Centers o /ID# 203292, Billings, Montana
  - Duplicate_Dartmouth-Hitchcock Medical Center - 1 Medical Center Drive /ID# 203350, Lebanon, New Hampshire
  - Titan Health Partners LLC, d/b/a Astera Cancer Care /ID# 228868, East Brunswick, New Jersey
  - Atlantic Health System /ID# 203404, Morristown, New Jersey
  - Capital Health Medical Center /ID# 203403, Pennington, New Jersey
  - Overlook Medical Center /ID# 211160, Summit, New Jersey
  - University of New Mexico /ID# 208339, Albuquerque, New Mexico
  - Duplicate_Gabrail Cancer Center Research /ID# 216056, Canton, Ohio
  - Univ Hosp Cleveland /ID# 215648, Cleveland, Ohio
  - Mercy Cancer Center /ID# 231972, Elyria, Ohio
  - Mercy Research Mercy Clinic Oklahoma Communities, Inc. / OKC /ID# 230154, Oklahoma City, Oklahoma
  - Providence Cancer Center Oncology and Hematology Care - Westside Portland /ID# 203301, Portland, Oregon
  - Penn State University and Milton S. Hershey Medical Center /ID# 221844, Hershey, Pennsylvania
  - Duplicate_Allegheny General Hospital /ID# 215585, Pittsburgh, Pennsylvania
  - Veterans Healthcare System /ID# 215602, Pittsburgh, Pennsylvania
  - Thompson Cancer Survival Ctr /ID# 228874, Knoxville, Tennessee
  - Vanderbilt Ingram Cancer Center /ID# 203281, Nashville, Tennessee
  - Houston Methodist Hospital /ID# 213268, Houston, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 216578, Temple, Texas
  - Virginia Cancer Specialists - Fairfax /ID# 203224, Fairfax, Virginia
  - Valley Medical Center /ID# 231459, Renton, Washington
  - University of Washington /ID# 206056, Seattle, Washington
  - Wisconsin Medical Center /ID# 210062, Milwaukee, Wisconsin
- Australia (5):
  - The Kinghorn Cancer Centre /ID# 207666, Darlinghurst, New South Wales
  - Newcastle Private Hospital /ID# 206600, Lambton Heights, New South Wales
  - The Tweed Hospital /ID# 206601, Tweed Heads, New South Wales
  - Mater Misericordiae Limited /ID# 229639, South Brisbane, Queensland
  - St John Of God Subiaco Hospital /ID# 226943, Subiaco, Western Australia
- Belgium (9):
  - Universitair Ziekenhuis Antwerpen /ID# 217430, Edegem, Antwerpen
  - Hospital La Louviere Site Jolimont - Helora /ID# 230586, La Louvière, Hainaut
  - Jessa Ziekenhuis /ID# 234047, Hasselt, Limburg
  - Vitaz /Id# 239966, Sint-Niklaas, Oost-Vlaanderen
  - Institut Jules Bordet /ID# 238614, Anderlecht
  - AZ Maria Middelares /ID# 233474, Ghent
  - AZ Groeninge /ID# 217431, Kortrijk
  - Duplicate_CHU de Liege /ID# 230589, Liège
  - UCL Namur University Hospital, Site Sainte-Elisabeth /ID# 234048, Namur
- Bulgaria (4):
  - MHAT Dobrich /ID# 230074, Dobrich
  - UMHAT Dr Georgi Stranski EAD /ID# 232024, Pleven
  - Medical Center Nadezhda /ID# 230473, Sofia
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 232010, Sofia
- Canada (4):
  - Duplicate_Cross Cancer Institute /ID# 204540, Edmonton, Alberta
  - Ottawa Hospital Research Institute /ID# 205579, Ottawa, Ontario
  - University Health Network_Princess Margaret Cancer Centre /ID# 204423, Toronto, Ontario
  - CISSS de la Monteregie /ID# 211356, Greenfield Park, Quebec
- China (20):
  - Anhui Provincial Hospital /ID# 212096, Hefei, Anhui
  - Anhui Provincial Cancer Hospital /ID# 239058, Hefei, Anhui
  - Anhui Medical University - Anhui Chest Hospital /ID# 239048, Hefei, Anhui
  - Beijing Cancer Hospital /ID# 210133, Beijing, Beijing Municipality
  - Fujian Provincial Cancer Hospital /ID# 210808, Fuzhou, Fujian
  - The First Affiliated Hospital Of Guangzhou Medical University /ID# 232261, Guangzhou, Guangdong
  - Affiliated Cancer Hospital of Guangxi Medical University /ID# 231560, Nanning, Guangxi
  - Affiliated Hospital of Hebei University /ID# 227262, Baoding, Hebei
  - Harbin Medical University Cancer Hospital /Id# 231573, Harbin, Heilongjiang
  - Henan Cancer Hospital /ID# 210961, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 211119, Wuhan, Hubei
  - The First People's Hospital of Changzhou /ID# 210787, Changzhou, Jiangsu
  - Jilin Cancer Hospital /ID# 210563, Changchun, Jilin
  - Shandong Cancer Hospital /ID# 231577, Jinan, Shandong
  - Shanghai Chest Hospital /ID# 210930, Shanghai, Shanghai Municipality
  - Fudan University Cancer Hospital /ID# 210084, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 210022, Chengdu, Sichuan
  - The Affiliated Cancer Hospital of Xinjiang Medical University /ID# 227244, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 211154, Hangzhou, Zhejiang
  - Zhejiang Cancer hospital /ID# 210085, Hangzhou, Zhejiang
- Czechia (2):
  - Duplicate_Vseobecna fakultni nemocnice v Praze /ID# 229797, Prague, Praha 17
  - Multiscan s.r.o. /ID# 241926, Prague
- France (10):
  - APHM - Hopital Nord /ID# 209854, Marseille, Bouches-du-Rhone
  - Institut Bergonie /ID# 216207, Bordeaux, Gironde
  - CHU Lille - Hôpital Albert Calmette /ID# 205105, Lille, Hauts-de-France
  - Institut Curie /ID# 207046, Paris, Paris
  - Hospices Civils de Lyon (HCL) - Hopital Louis Pradel /ID# 216209, Bron, Rhone
  - Centre Leon Berard /ID# 205107, Lyon, Rhone
  - Centre Hosp Intercommunal de Creteil /ID# 227108, Créteil, Val-de-Marne
  - Institut Gustave Roussy /ID# 205149, Villejuif, Val-de-Marne
  - CHI Toulon-La Seyne sur Mer /ID# 230545, Toulon, Var
  - CHU Strasbourg - Hopital Civil /ID# 208080, Strasbourg
- Germany (9):
  - Universitatsklinikum Mannheim /ID# 228798, Mannheim, Baden-Wurttemberg
  - Gemeinschaftspraxis Dr. Heinrich und Prof. Bangerter /ID# 232052, Augsburg, Bavaria
  - Universitaetsklinikum Giessen /ID# 231856, Giessen, Hesse
  - Klinikum Kassel /ID# 205443, Kassel, Hesse
  - Pius-Hospital Oldenburg /ID# 211615, Oldenburg, Lower Saxony
  - Krankenhaus Martha-Maria Halle-Doelau /ID# 205442, Halle, Saxony-Anhalt
  - Vivantes Klinikum Neukolln /ID# 205928, Berlin
  - Asklepios Fachkliniken Muenchen-Gauting /ID# 207789, Gauting
  - Evangelisches Krankenhaus Hamm /ID# 208043, Hamm
- Greece (5):
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 205528, Athens, Attica
  - Metropolitan Hospital /ID# 205529, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 205530, Heraklion, Crete
  - Bioclinic Thessaloniki /ID# 227261, Thessaloniki
  - Euromedica General Clinic /ID# 227264, Thessaloniki
- Hungary (5):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 204878, Encs, Borsod-Abauj Zemplen county
  - Torokbalinti Tudogyogyintezet /ID# 204883, Törökbálint, Pest County
  - Duplicate_Semmelweis Egyetem /ID# 204434, Budapest
  - Duplicate_Veszprem Megyei Tudogyogyintez /ID# 213950, Farkasgyepű
  - Matrai Gyogyintezet /ID# 204432, Mátraháza
- Ireland (4):
  - Cork University Hospital /ID# 205103, Wilton, Cork
  - Mater Misericordiae Univ Hospital /ID# 231466, Dublin, Dublin
  - St James Hospital /ID# 205104, Dublin, Dublin
  - St Vincents University Hospital /ID# 205102, Elm Park, Dublin
- Israel (5):
  - Meir Medical Center /ID# 204255, Kfar Saba, Central District
  - Soroka University Medical Center /ID# 204898, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 204254, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 204866, Haifa
  - Rabin Medical Center /ID# 215322, Petah Tikva
- Italy (10):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 216153, Bologna, Emilia-Romagna
  - Duplicate_Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRCCS /ID# 205601, Meldola, Forlì-Cesena
  - IRCCS Ospedale San Raffaele /ID# 226973, Milan, Milano
  - Azienda Ospedaliera Universitaria Federico II /ID# 231948, Naples, Napoli
  - Duplicate_IRCCS Istituti Fisioterapici Ospitalieri-Istituto Nazionale Tumori Reg /ID# 227011, Rome, Roma
  - Azienda Ospedaliera San Camillo Forlanini /ID# 205163, Rome, Roma
  - Duplicate_A.O.U. San Luigi Gonzaga /ID# 204706, Orbassano, Torino
  - L'Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialità San Giuseppe Mos /ID# 204707, Avellino
  - Azienda Ospedaliero-Universitaria di Parma /ID# 204983, Parma
  - Fondazione Policlinico Universitario Campus Bio-Medico /ID# 215918, Roma
- Japan (27):
  - Chukyo Hospital /ID# 244755, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 207790, Nagoya, Aichi-ken
  - Hirosaki University Hospital /ID# 245023, Hirosaki-shi, Aomori
  - Duplicate_Chiba University Hospital /ID# 232204, Chiba, Chiba
  - Duplicate_National Hospital Organization Shikoku Cancer Center /ID# 232252, Matsuyama, Ehime
  - Duplicate_National Hospital Organization Kyushu Cancer Center /ID# 206061, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 227776, Kurume-shi, Fukuoka
  - Chugoku Central Hospital /ID# 245022, Fukuyama, Hiroshima
  - Hiroshima Citizens Hospital /ID# 218087, Hiroshima, Hiroshima
  - Himeji Medical Center /ID# 227777, Himeji-shi, Hyōgo
  - Kobe Minimally Invasive Cancer Center /ID# 248590, Kobe, Hyōgo
  - Takarazuka City Hospital /ID# 245185, Takarazuka-shi, Hyōgo
  - Yokohama Municipal Citizen's Hospital /ID# 248374, Yokohama, Kanagawa
  - Duplicate_Kanagawa Cancer Center /ID# 205068, Yokohama, Kanagawa
  - Matsusaka Municipal Hospital /ID# 230219, Matsusaka-shi, Mie-ken
  - Sendai Kousei Hospital /ID# 216460, Sendai, Miyagi
  - Niigata Cancer Center Hospital /ID# 216462, Niigata, Niigata
  - Okayama University Hospital /ID# 227851, Okayama, Okayama-ken
  - Osaka City General Hospital /ID# 233172, Osaka, Osaka
  - Osaka International Cancer Institute /ID# 210735, Osaka, Osaka
  - NHO Kinki Chuo Chest Medical Center /ID# 216461, Sakai-shi, Osaka
  - Duplicate_Saitama Cancer Center /ID# 232508, Kitaadachi-gun, Saitama
  - Fujieda Municipal General Hospital /ID# 248589, Fujieda-shi, Shizuoka
  - Duplicate_Duplicate_Duplicate_Shizuoka Cancer Center /ID# 205065, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 205066, Chuo-ku, Tokyo
  - Duplicate_The Cancer Institute Hospital Of JFCR /ID# 216463, Koto-ku, Tokyo
  - Yamaguchi - Ube Medical Center /ID# 227778, Ube-shi, Yamaguchi
- Netherlands (3):
  - Ziekenhuis St. Jansdal /ID# 216658, Harderwijk, Gelderland
  - Antoni van Leeuwenhoek /ID# 216657, Amsterdam, North Holland
  - Meander Medisch Centrum /ID# 217756, Amersfoort, Utrecht
- Poland (5):
  - Med Polonia Sp. z o. o. /ID# 229908, Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Bada /ID# 230595, Warsaw, Masovian Voivodeship
  - Wojewodzki Szpital im. Sw. Ojca Pio /ID# 231960, Przemyśl, Podkarpackie Voivodeship
  - Dom Lekarski S.A. /ID# 231479, Szczecin, West Pomeranian Voivodeship
  - Duplicate_Uniwersytecki Szpital Kliniczny im. Wojskowej Akademii Medycznej /ID# 231476, Lodz, Łódź Voivodeship
- Puerto Rico (2):
  - VA Caribbean Healthcare System /ID# 206336, San Juan
  - Puerto Rico Hematology Oncolog /ID# 206337, San Juan
- Romania (7):
  - Institutul Oncologic Prof Dr. Ion Chiricuta Cluj Napoca /ID# 206320, Cluj-Napoca, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie S.R.L. /ID# 227623, Craiova, Dolj
  - Spitalul Municipal Ploiesti /ID# 229097, Ploieşti, Prahova
  - Oncomed SRL /ID# 205616, Timișoara, Timiș County
  - Institutul Oncologic Prof. Dr. Alexandru Trestioreanu Bucuresti /ID# 227216, Bucharest
  - Spitalul Clinic Coltea /ID# 227241, Bucharest
  - S.C. Gral Medical Srl /Id# 227215, Bucharest
- Russia (15):
  - Krasnoyarsk Regional Clinical Oncology Dispensary n.a. A.I. Kryzhanovsky /ID# 232065, Krasnoyarsk, Krasnoyarsk Krai
  - LLC Medical Center /ID# 212397, Novosibirsk, Novosibirsk Oblast
  - Clinical Oncology Dispensary of Omsk /ID# 239313, Omsk, Omsk Oblast
  - St. Petersburg scientific center for specialized medical care (oncological) /ID# 206405, Saint Petersburg, Sankt-Peterburg
  - Newclinic Medical Center /ID# 216262, Pyatigorsk, Stavropol Kray
  - Republican Clinical Oncology Dispensary /ID# 206463, Kazan', Tatarstan, Respublika
  - Regional Children's Clinical Hospital of Volgograd /ID# 206520, Volgograd, Volgograd Oblast
  - Arkhangelsk Clinical Oncology Dispensary /ID# 216418, Arkhangelsk
  - Evimed Clinic /ID# 216473, Chelyabinsk
  - Kostroma region oncology center /ID# 231317, Kostroma
  - Univercity Headache Clynic,LTD /ID# 212080, Moscow
  - VitaMed LLC /ID# 228957, Moscow
  - National Medical Research Radiological Centre /ID# 231263, Obninsk
  - Euromedservice /ID# 206390, Pushkin
  - Center of Palliative Medicine De Vita /ID# 212900, Saint Petersburg
- South Korea (9):
  - National Cancer Center /ID# 204241, Goyang-si, Gyeonggido
  - Duplicate_Seoul National University Bundang Hospital /ID# 204237, Seongnam, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 229647, Suwon, Gyeonggido
  - Pusan National University Yangsan Hospital /ID# 233871, Yangsan, Gyeongsangnam-do
  - Inha University Hospital /ID# 234206, Incheon, Incheon Gwang Yeogsi
  - Chonnam National University Hwasun Hospital /ID# 206951, Hwasun-gun, Jeonranamdo
  - Duplicate_Chungbuk National Univ Hosp /ID# 205680, Cheongju-si, North Chungcheong
  - Asan Medical Center /ID# 204236, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 227083, Seoul, Seoul Teugbyeolsi
- Spain (13):
  - Duplicate_Hospital Clínico Universitario de Santiago-CHUS /ID# 204367, Santiago de Compostela, A Coruna
  - Instituto Catalan de Oncologia (ICO) Badalona /ID# 216106, Badalona, Barcelona
  - CHU Insular-Materno Infantil /ID# 232362, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Fundacion Alcorcon /ID# 232361, Alcorcón, Madrid
  - Hospital Nuestra Senora de Sonsoles /ID# 232367, Ávila
  - Hospital Universitario Dexeus - Grupo Quironsalud /ID# 232368, Barcelona
  - Hospital Universitario Vall de Hebron /ID# 206997, Barcelona
  - Hospital Universitario Ramon y Cajal /ID# 203922, Madrid
  - Hospital Universitario HM Sanchinarro /ID# 203913, Madrid
  - Hospital Regional Universitario de Malaga /ID# 216081, Málaga
  - Hospital Universitario Virgen Macarena /ID# 230998, Seville
  - Hospital Universitario Virgen del Rocio /ID# 216058, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 203862, Valencia
- Switzerland (2):
  - University Hospital Basel /ID# 230977, Basel Town, Canton of Basel-City
  - KSW Kantonsspital Winterthur /ID# 231284, Winterthur, Canton of Zurich
- Taiwan (9):
  - Duplicate_Kaohsiung Chang Gung Memorial Hospital /ID# 205423, Kaohsiung City, Kaohsiung
  - National Taiwan University Hospital /ID# 205100, Taipei City, Taipei
  - Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation /ID# 205309, Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 205831, Kaohsiung City
  - Taipei Medical University Shuang Ho Hospital /ID# 215356, New Taipei City
  - Taichung Veterans General Hospital /ID# 205308, Taichung
  - National Cheng Kung University Hospital /ID# 205307, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center /ID# 227336, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 205424, Taoyuan
- Turkey (Türkiye) (7):
  - Adana Sehir Egitim ve Arastirma Hastanesi /ID# 206000, Adana
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi /ID# 205243, Ankara
  - Gazi University Medical Faculty /ID# 239816, Ankara
  - Akdeniz Universitesi Tip Fakul /ID# 205238, Antalya
  - Trakya University Medical Facu /ID# 205242, Edirne, Istanbul
  - Prof. Dr. Suleyman Yalcın Sehir Hastanesi /ID# 215082, Istanbul
  - Dr. Suat Seren Gogus Has /ID# 215083, Izmir
- United Kingdom (5):
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 239889, London, Greater London
  - University College London Hospital /ID# 231467, London, Greater London
  - Nottingham City Hospital /ID# 231224, Nottingham, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust /ID# 205890, Oxford, Oxfordshire
  - University Hospitals Birmingham NHS Foundation Trust /ID# 206209, Birmingham

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Camidge DR, Bar J, Horinouchi H, Goldman J, Moiseenko F, Filippova E, Cicin I, Ciuleanu T, Daaboul N, Liu C, Bradbury P, Moskovitz M, Katgi N, Tomasini P, Zer A, Girard N, Cuppens K, Han JY, Wu SY, Baijal S, Mansfield AS, Kuo CH, Nishino K, Lee SH, Planchard D, Baik C, Li M, Ansell P, Xia S, Bolotin E, Looman J, Ratajczak C, Lu S. Telisotuzumab Vedotin Monotherapy in Patients With Previously Treated c-Met Protein-Overexpressing Advanced Nonsquamous EGFR-Wildtype Non-Small Cell Lung Cancer in the Phase II LUMINOSITY Trial. J Clin Oncol. 2024 Sep 1;42(25):3000-3011. doi: 10.1200/JCO.24.00720. Epub 2024 Jun 6. PMID 38843488